CLINICAL TRIAL: NCT01003106
Title: RanibizumabDosE Comparison (0.5mg and 2.0mg) and the Role of LAser in the ManagemenT of REtinal Vein Occlusion - A Pharmacodynamic Approach(RELATE)
Brief Title: Ranibizumab DosE Comparison and the Role of LAser in REtinal Vein Occlusions
Acronym: RELATE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter A Campochiaro, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Peter A Campochiaro, MD, Principal Investigator, Johns Hopkins University
Organization: Johns Hopkins University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00032394
Record Dates: First submitted 2009-10-26; First posted 2009-10-28 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Retinal Vein Occlusion
Keywords: RVO; BRVO; CRVO; Vein occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- BRVO- Ranibizumab 0.5mg alone (Experimental): Branch retinal vein occlusion patients randomized to this group will receive 0.5mg of ranibizumab alone as per protocol without laser photocoagulation.
  Interventions: Drug: Ranibizumab 0.5mg (monthly)
- BRVO- Pro re nata (prn) ranibizumab with laser (Experimental): Branch retinal vein occlusion patients randomized to this group will receive 0.5mg/2.0mg of ranibizumab as per protocol, and additional laser photocoagulation if required.
  Interventions: Drug: Pro re nata (prn) ranibizumab; Procedure: Pro re nata (prn) Laser photocoagulation
- BRVO- Ranibizumab 2.0mg alone (Experimental): Branch retinal vein occlusion patients randomized to this group will receive 2.0mg of ranibizumab alone as per protocol without laser photocoagulation.
  Interventions: Drug: Ranibizumab 2.0mg (monthly)
- BRVO- Pro re nata (prn) ranibizumab (Experimental): Branch retinal vein occlusion patients randomized to this group will receive 0.5mg/2.0mg of ranibizumab as per protocol, without additional laser photocoagulation.
  Interventions: Drug: Pro re nata (prn) ranibizumab
- CRVO- Ranibizumab 0.5mg alone (Experimental): Central retinal vein occlusion patients randomized to this group will receive 0.5mg of ranibizumab alone as per protocol without laser photocoagulation
  Interventions: Drug: Ranibizumab 0.5mg (monthly)
- CRVO- Pro re nata (prn) ranibizumab with laser (Experimental): Central retinal vein occlusion patients randomized to this group will receive 0.5mg/2.0mg of ranibizumab as per protocol, and additional laser photocoagulation if required.
  Interventions: Drug: Pro re nata (prn) ranibizumab; Procedure: Pro re nata (prn) Laser photocoagulation
- CRVO- Ranibizumab 2.0mg alone (Experimental): Central retinal vein occlusion patients randomized to this group will receive 2.0mg of ranibizumab alone as per protocol without laser photocoagulation.
  Interventions: Drug: Ranibizumab 2.0mg (monthly)
- CRVO- Pro re nata (prn) ranibizumab (Experimental): Central retinal vein occlusion patients randomized to this group will receive 0.5mg/2.0mg of ranibizumab as per protocol, without additional laser photocoagulation.
  Interventions: Drug: Pro re nata (prn) ranibizumab

INTERVENTIONS:
Drug: Ranibizumab 0.5mg (monthly) — Branch retinal vein occlusion- Intravitreal injection of 0.5mg ranibizumab alone
  Arms: BRVO- Ranibizumab 0.5mg alone; CRVO- Ranibizumab 0.5mg alone
Drug: Ranibizumab 2.0mg (monthly)
  Arms: BRVO- Ranibizumab 2.0mg alone; CRVO- Ranibizumab 2.0mg alone
Drug: Pro re nata (prn) ranibizumab
  Arms: BRVO- Pro re nata (prn) ranibizumab; BRVO- Pro re nata (prn) ranibizumab with laser; CRVO- Pro re nata (prn) ranibizumab; CRVO- Pro re nata (prn) ranibizumab with laser
Procedure: Pro re nata (prn) Laser photocoagulation
  Arms: BRVO- Pro re nata (prn) ranibizumab with laser; CRVO- Pro re nata (prn) ranibizumab with laser

SUMMARY:
The primary Objective of this study is to evaluate the safety and tolerability of intraocular injections of 0.5mg or 2.0mg of ranibizumab in patients with macular edema due to retinal vein occlusion.

DETAILED DESCRIPTION:
The secondary objectives are to assess the efficacy of 0.5mg versus 2.0mg of monthly ranibizumab injections in patients with macular edema due to retinal vein occlusion between baseline and month 6. At week 24, patients will be re-randomized to receive pro re nata (prn) ranibizumab+laser photocoagulation versus ranibizumab alone and the efficacy of both treatment options will be compared. Treatment efficacy will be assessed by comparing changes in best corrected visual acuity (BCVA) and central subfiled thickness (CST) between the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age equal to or greater than 18 years
* Diagnosis of macular edema due to central or branch retinal vein occlusion
* Foveal thickness of equal to or greater than 250 mm, as assessed by OCT
* Best corrected visual acuity score in the study eye of 20/40 to 20/400 inclusive (Snellen equivalents using the ETDRS protocol at a distance of 4 meters). Only one eye will be treated in the study. If both eyes are eligible, the investigator will select the eye to be enrolled.
* In the opinion of the investigator, decreased vision in the study eye is due to foveal thickening from vein occlusion and not from other obvious causes of decreased vision

Exclusion Criteria:

* Scatter laser photocoagulation or macular photocoagulation within 3 months of study entry in the study eye
* Intraocular surgery in the study eye within 3 months of study entry
* Use of intraocular or periocular injection of steroids in the study eye (e.g., triamcinolone) within 4 months of study entry
* Previous use of an anti-VEGF drug within 3 months of study entry
* Cataract surgery in the study eye within 3 months of study entry; Yttrium-Aluminum-Garnet (YAG) laser capsulotomy within 1 month of study entry; or any other intraocular surgery within 3 months preceding Day 0.
* History of vitreoretinal surgery in the study eye within 3 months of study entry
* Uncontrolled glaucoma (defined as intraocular pressure ³30 mm Hg despite treatment with anti-glaucoma medications)
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 3 months of study enrollment.
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Have the presence of active malignancy, including lymphoproliferative disorders. Subjects with a history of fully resolved basal or squamous cell skin cancer may be enrolled.
* Any condition that the investigator believes would pose a significant hazard to the subject if investigational therapy were initiated.
* History of allergy to humanized antibodies or any component of the ranibizumab formulation
* Inability to comply with study or followup procedures
* Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute at Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty-one patients with retinal vein occlusion were enrolled at a single center (The Wilmer Eye Institute, Johns Hopkins Hospital, Baltimore,MD).
Groups:
- BRVO- Ranibizumab 0.5mg Alone: Branch retinal vein occlusion patients randomized to this group at baseline will receive 0.5mg of ranibizumab alone for 6 months.
- BRVO- Ranibizumab 2.0mg Alone: Branch retinal vein occlusion patients randomized to this group at baseline will receive 2.0mg of Ranibizumab alone for 6 months.
- BRVO- Pro re Nata (Prn) Ranibizumab Alone: Branch retinal vein occlusion patients randomized to this group at month 6 will receive pro re nata 0.5mg/2.0mg of ranibizumab without laser photocoagulation.
- BRVO- Pro re Nata (Prn) Ranibizumab+Laser Photocoagulation: Branch retinal vein occlusion patients randomized to this group at month 6 will receive pro re nata (prn) ranibizumab along with laser photocoagulation.
- CRVO- Ranibizumab 0.5mg Alone: Central retinal vein occlusion patients randomized to this group at baseline will receive 0.5mg at of ranibizumab alone for 6 months.
- CRVO- Ranibizumab 2.0mg Alone: Central retinal vein occlusion patients randomized to this group at baseline will receive ranibizumab 2.0mg alone for 6 months .
- CRVO- Pro re Nata (Prn) Ranibizumab Alone: Central retinal vein occlusion patients randomized to this group at month 6 will receive pro re nata (prn) 0.5mg/2.0mg ranibizumab alone without laser photocoagulation.
- CRVO- Pro re Nata (PRN) Ranibizumab+Laser Photocoagulation: Central retinal vein occlusion patients randomized to this group at month 6 will receive 0.5mg/2.0mg prn ranibizumab along with laser photocoagulation.
Period: Baseline to Month 6
Arm/Group | BRVO- Ranibizumab 0.5mg Alone | BRVO- Ranibizumab 2.0mg Alone | BRVO- Pro re Nata (Prn) Ranibizumab Alone | BRVO- Pro re Nata (Prn) Ranibizumab+Laser Photocoagulation | CRVO- Ranibizumab 0.5mg Alone | CRVO- Ranibizumab 2.0mg Alone | CRVO- Pro re Nata (Prn) Ranibizumab Alone | CRVO- Pro re Nata (PRN) Ranibizumab+Laser Photocoagulation
Started | 22 | 20 | 0 | 0 | 19 | 20 | 0 | 0
Completed | 22 | 20 | 0 | 0 | 19 | 20 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Month 6-Month 36
Arm/Group | BRVO- Ranibizumab 0.5mg Alone | BRVO- Ranibizumab 2.0mg Alone | BRVO- Pro re Nata (Prn) Ranibizumab Alone | BRVO- Pro re Nata (Prn) Ranibizumab+Laser Photocoagulation | CRVO- Ranibizumab 0.5mg Alone | CRVO- Ranibizumab 2.0mg Alone | CRVO- Pro re Nata (Prn) Ranibizumab Alone | CRVO- Pro re Nata (PRN) Ranibizumab+Laser Photocoagulation
Started | 0 | 0 | 19 | 20 | 0 | 0 | 20 | 18
Completed | 0 | 0 | 18 | 20 | 0 | 0 | 19 | 18
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- BRVO- Ranibizumab 0.5mg Alone: Branch retinal vein occlusion patients randomized to this group will receive 0.5mg of ranibizumab alone as per protocol without laser photocoagulation.
  BRVO -Ranibizumab 0.5mg alone: Branch retinal vein occlusion- Intravitreal injection of 0.5mg ranibizumab alone
- BRVO- Ranibizumab 2.0mg Alone: Branch retinal vein occlusion patients randomized to this group will receive 2.0mg of ranibizumab alone as per protocol without laser photocoagulation.
  BRVO- Ranibizumab 2.0 mg alone: Branch retinal vein occlusion- Intravitreal injection of 2.0mg ranibizumab alone
- CRVO- Ranibizumab 0.5mg Alone: Central retinal vein occlusion patients randomized to this group will receive 0.5mg of ranibizumab alone as per protocol without laser photocoagulation
  CRVO -Ranibizumab 0.5mg alone: Central retinal vein occlusion- Intravitreal injection of 0.5mg ranibizumab alone
- CRVO- Ranibizumab 2.0mg Alone: Central retinal vein occlusion patients randomized to this group will receive 2.0mg of ranibizumab alone as per protocol without laser photocoagulation.
  CRVO- Ranibizumab 2.0 mg alone: Central retinal vein occlusion- Intravitreal injection of 2.0mg ranibizumab alone
- Total: Total of all reporting groups
Arm/Group | BRVO- Ranibizumab 0.5mg Alone | BRVO- Ranibizumab 2.0mg Alone | CRVO- Ranibizumab 0.5mg Alone | CRVO- Ranibizumab 2.0mg Alone | Total
Number analyzed (Participants) | 22 | 20 | 19 | 20 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (2.2) | 69.3 (1.8) | 59.0 (2.9) | 64.4 (2.9) | 64.7 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 9 | 9 | 38
  Male | 9 | 13 | 10 | 11 | 43

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Ocular and Non-ocular Adverse Events.
Time Frame: 36 months
Measure: Number; unit: participants
Groups:
- BRVO: Patients with Branch Retinal Vein Occlusion
- CRVO: Patients with Central Retinal Vein Occlusion
Arm/Group | BRVO | CRVO
Number analyzed (Participants) | 42 | 39
participants
  Patients with Serious Adverse Events | 17 | 12
  Patient with (non serious) adverse events | 37 | 35

2. Secondary Outcome: Mean Change From Baseline to Month 6 in Best Corrected Visual Acuity in Patients Treated With 0.5mg Versus 2.0mg of Ranibizumab
Time Frame: Baseline to month 6
Measure: Mean (Standard Error); unit: Letters
Groups:
- BRVO-Ranibizumab 0.5mg Alone: Branch retinal vein occlusion patients randomized to this group will receive 0.5mg of ranibizumab alone.
- BRVO- Ranibizumab 2.0mg Alone: Branch retinal vein occlusion patients randomized to this group will receive 2.0mg of ranibizumab alone.
- CRVO- Ranibizumab 0.5mg Alone: Patients randomized to receive 0.5mg of ranibizumab alone
- CRVO- Ranibizumab 2.0mg Alone: Central retinal vein occlusion patients randomized to receive 2.0mg of ranibizumab alone.
Arm/Group | BRVO-Ranibizumab 0.5mg Alone | BRVO- Ranibizumab 2.0mg Alone | CRVO- Ranibizumab 0.5mg Alone | CRVO- Ranibizumab 2.0mg Alone
Number analyzed (Participants) | 22 | 20 | 19 | 20
Letters | 12.1 (2.9) | 14.6 (2.3) | 15.5 (2.4) | 15.8 (2.4)

3. Secondary Outcome: Mean Change From Month 6 to Month 36 in Best Corrected Visual Acuity in Patients Treated With Prn Ranibizumab+Laser Photocoagulation Versus Prn Ranibizumab Alone.
Time Frame: Month 6- Month 36
Measure: Mean (Standard Error); unit: Letters
Groups:
- BRVO- Pro re Nata (Prn) Ranibizumab Alone: Branch retinal vein occlusion patients in this group will receive pro re nata 0.5mg/2.0mg of ranibizumab along without laser photocoagulation.
- BRVO- Pro re Nata (Prn) Ranibizumab+Laser Photocoagulation: Branch retinal vein occlusion patients in this group will receive pro re nata (prn) ranibizumab and laser.
- CRVO- Pro re Nata (Prn) Ranibizumab Alone: Central retinal vein occlusion patients in this group will receive pro re nata (prn) 0.5mg/2.0mg ranibizumab alone without laser photocoagulation.
- CRVO- Pro re Nata (PRN) Ranibizumab+Laser Photocoagulation: Central retinal vein occlusion patients in this group will receive 0.5mg/2.0mg prn ranibizumab and laser photocoagulation.
Arm/Group | BRVO- Pro re Nata (Prn) Ranibizumab Alone | BRVO- Pro re Nata (Prn) Ranibizumab+Laser Photocoagulation | CRVO- Pro re Nata (Prn) Ranibizumab Alone | CRVO- Pro re Nata (PRN) Ranibizumab+Laser Photocoagulation
Number analyzed (Participants) | 18 | 20 | 19 | 18
Letters | 3.1 (3.3) | -2.6 (2.2) | -6.7 (3.7) | 0.4 (4.3)

4. Secondary Outcome: Mean Change From Baseline to Month 6 in Central Subfield Thickness in Patients Treated With 0.5mg Versus 2.0mg of Ranibizumab
Time Frame: Baseline to month 6
Measure: Mean (Standard Error); unit: microns
Arm/Group | BRVO-Ranibizumab 0.5mg Alone | BRVO- Ranibizumab 2.0mg Alone | CRVO- Ranibizumab 0.5mg Alone | CRVO- Ranibizumab 2.0mg Alone
Number analyzed (Participants) | 22 | 20 | 19 | 20
microns | -203.3 (41) | -292.1 (55) | -253.5 (43) | -396.1 (48.1)

5. Secondary Outcome: Mean Change From Month 6 to Month 36 in Central Subfield Thickness in Patients Treated With Prn Ranibizumab+Laser Photocoagulation Versus Prn Ranibizumab Alone.
Time Frame: Month 6- Month 36
Measure: Mean (Standard Error); unit: microns
Arm/Group | BRVO- Pro re Nata (Prn) Ranibizumab Alone | BRVO- Pro re Nata (Prn) Ranibizumab+Laser Photocoagulation | CRVO- Pro re Nata (Prn) Ranibizumab Alone | CRVO- Pro re Nata (PRN) Ranibizumab+Laser Photocoagulation
Number analyzed (Participants) | 18 | 20 | 19 | 18
microns | -3.2 (54.7) | 36.6 (29.2) | 19.1 (50.3) | 58.8 (38.5)

ADVERSE EVENTS:
Time Frame: From Baseline to Month 36
Arm/Group | BRVO | CRVO
Serious Adverse Events (participants affected / at risk) | 17/42 | 12/39
Other Adverse Events (participants affected / at risk) | 37/42 | 35/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRVO (N=42) | CRVO (N=39)
Urinary Tract Infection Requiring Hospitalization (Renal and urinary disorders) | 1 (1) | 0 (0)
Worsening of Cataract/Cataract Surgery (Eye disorders) | 3 (3) | 2 (2)
Hospitalization for Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Vertebral Fracture/Surgery (Surgical and medical procedures) | 2 (2) | 1 (1)
Cerebrovascular event (Nervous system disorders) | 2 (2) | 0 (0)
Hospitalization for Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Knee surgery (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Vitreous Hemorrhage resulting in significant visual loss (Eye disorders) | 1 (1) | 1 (1)
Severe Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Kidney Surgery (Renal and urinary disorders) | 1 (1) | 0 (0)
Trabulectomy (Eye disorders) | 1 (1) | 0 (0)
Severe Cheat pain/Acute Coronary Syndrome (Cardiac disorders) | 2 (2) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Colon Surgery (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hospitalization due to multiple systemic diseases (General disorders) | 1 (1) | 1 (1)
Brain Surgery (Nervous system disorders) | 1 (1) | 0 (0)
Transient global Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Serious Drug Allergy requiring Hospitalization (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertensive Crisis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Surgery for Macular Pucker (Eye disorders) | 0 (0) | 1 (1)
Hospitalization for Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Parotid Gland Swelling (Endocrine disorders) | 0 (0) | 1 (1)
Pancreatic Mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRVO (N=42) | CRVO (N=39)
Increased IOP (Eye disorders) | 2 (2) | 0 (0)
Tooth Extraction (General disorders) | 3 (3) | 0 (0)
Skin Lesion/Skin Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Headache (General disorders) | 2 (2) | 0 (0)
Common Cold/cough (General disorders) | 10 (10) | 10 (10)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Sinusitis (General disorders) | 2 (2) | 3 (3)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Worsening Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Hernia Repair Surgery (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fall (General disorders) | 2 (2) | 0 (0)
Back Pain (General disorders) | 5 (5) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 7 (7) | 7 (7)
Blurry vision (Eye disorders) | 0 (0) | 4 (4)
Vitreous Hemorrhage (Eye disorders) | 0 (0) | 2 (2)
Squamous Cell/Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Worsening Hypercholesterlemia (General disorders) | 0 (0) | 2 (2)
Foot Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Seasonal Allergy (General disorders) | 0 (0) | 3 (3)
Gout (General disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No